CLINICAL TRIAL: NCT06665763
Title: The Lactate Project: Investigating the Impact of Lactate to Preserve Vital Organ Blood Supply and Function in Heart and Brain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: THE LACTATE PROJECT
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Lactate Blood Increase
Keywords: Human metabolism; Substrate utilization; Cerebral blod flow; Cardiac metabolism; Cerebral metabolism; Cardiac perfusion; Glucose metabolism; Lipid metabolism; Lactate utilization
MeSH Terms: conditions — Hyperlactatemia

STUDY DESIGN:
Intervention Model Description: The study will be carried out as a single-blinded, randomized cross-over clinical investigational trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Na-Lactate infusion (Experimental)
  Interventions: Other: Sodium Lactate Solution
- Saline infusion (Placebo) (Placebo Comparator)
  Interventions: Other: Saline infusion (placebo)

INTERVENTIONS:
Other: Sodium Lactate Solution — Infusion of sodium-lactate solution
  Arms: Na-Lactate infusion
Other: Saline infusion (placebo) — NaCl solution
  Other Names: NaCl
  Arms: Saline infusion (Placebo)

SUMMARY:
The aim of the proposed study is to investigate the effect of increased plasma lactate concentrations on the heart and brain's metabolism of other energy sources, primarily glucose in the brain and glucose and FFA in the heart.

The investigator hypothesize that:

* An acute increase in lactate plasma concentration will decrease cerebral glucose uptake and increase cerebral blood flow
* An acute increase in lactate plasma concentration will decrease palmitate and glucose uptake in the myocardium, and increase myocardial perfusion

DETAILED DESCRIPTION:
SCREENING VISIT

During the initial screening visit, the investigators will inform all potential volunteers about the project, and volunteers will have the chance to ask questions about participation in the project.

The investigators will register the following data

1. Medical history to assess exclusion criteria
2. Weight, height, BMI
3. Standard medical examination including pulse, blood pressure and an ECG

After assessment of inclusion- and exclusion criteria remaining volunteers will be offered to participate in the project. The investigators will screen potential volunteers with the following blood samples: haemoglobin, HbA1c, glucose, cholesterol, triglyceride, TSH, creatinine, albumin, sodium, potassium, ALAT, ASAT, bilirubin and coagulation parameters.

Blood samples and randomization will not take place until volunteers have signed the informed consent form.

MAGNETIC RESONANCE IMAGING (MRI) SCAN

The investigators will perform a cerebral MRI for the purpose of anatomical localisation for alignment with the PET scans on the 1st and 2nd study day.

1st STUDY DAY:

The volunteers will arrive fasted (8 hours) at the Department of Nuclear Medicine & PET-Centre at 7.30 a.m., where the subject will have an arterial catheter placed for arterial blood sampling during PET scans as well as two venous catheters for blood sampling and continued administration of intravenous fluids (saline or Na-lactate) and adenosine. At 9.00 a.m., we will start the Na-lactate or saline infusion.

From 9.30 a.m., the investigators will perform PET scans with administration of relevant PET tracers preceding each scan. The investigators will perform PET scans in the following order:

1. Dynamic PET scan with [15O]H2O in order to assess cerebral perfusion.
2. Dynamic PET scan with [15O]H2O in order to assess myocardial perfusion.
3. Stress test using an adenosine infusion during a dynamic PET scan with [15O]H2O to assess coronary flow reserve (CFR) in the heart.
4. Dynamic PET scan with [11C]Palmitate to assess uptake, oxidation and re-esterification of FFA in the heart.
5. Dynamic PET scan with [11C]Acetate to asses oxygen and energy expenditure in the heart.
6. Dynamic whole-body PET scan with [18F]FDG to assess glucose uptake in the heart and brain.

Following the [11C]Acetate scan the investigators will administrate a continued infusion of insulin (0,3 mIE/kg/min) and 20% glucose throughout the rest of the study day in order to achieve hyperinsulinemic-euglycemic conditions (clamp conditions). To correct for attenuation, we will perform three lowdose, non-contrast enhanced CT scans over the course of the study day. The investigators will draw blood samples every hour.

2nd STUDY DAY

The PET scan regime during the 2nd study day is identical to the 1st study day. If volunteers were administered Na-lactate during the 1st study day they will be administered saline during the 2nd studyday and vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-75 years
2. Male or postmenopausal female
3. BMI 20-35 kg/m2
4. Signed informed consent form

Exclusion Criteria:

1. Clinically significant heart, lung, kidney, kidney, liver, endocrine or malignant disease basedon information obtained during an initial screening visit as well as blood samples and an ECG.
2. Blood donation within the last 3 months
3. Smoking
4. Alcohol- or substance abuse
5. Participation in other clinical trials involving ionized radiation within the last 6 months
6. Claustrophobia

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral glucose uptake | From T=300-360 (minutes)
  Cerebral glucose uptake ([18F]FDG PET scan) under basal and hyperinsulinemic- euglycemic conditions (clamp conditions).

SECONDARY OUTCOMES:
Cerebral blood flow | T = 0-10 (minutes)
  Cerebral blood flow ([15O]H2O PET scan)
Myocardial perfusion | T = 0-10 (minutes)
  Myocardial perfusion ([15O]H2O PET scan)
Myocardial glucose uptake | T = 300-360 (minutes)
  Myocardial glucose uptake ([18F]FDG PET scan)
Myocardial FFA uptake and oxidation | T = 30-70 (minutes)
  Myocardial FFA uptake and oxidation ([11C]Palmitate PET scan)
Myocardial contractility | T=0-10 (minutes)
  Myocardial contractility (ejection fraction based on ECG-gated PET scan)
Myocardial oxygen consumption and efficiency | T=150-180 (minutes)
  Myocardial oxygen consumption and efficiency ([11C]Acetate PET scan)
Blood sampling | T = -60 to 360 (minutes)
  A number of cardiometabolic blood samples will be collected during the whole study day.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Medical Research Laboratories/Steno Diabetes Center Aarhus, Aarhus, N
  - Department of Nuclear Medicine & PET-Centre, Aarhus, N

IPD SHARING:
Plan to Share IPD: No